CLINICAL TRIAL: NCT07241663
Title: Conversion Surgery for Locally Unresectable Pancreatic Cancer - International Multi-center Observational Trial (ROBIN= suRgery for lOcally unresectaBle pancreatIc Cancer)
Brief Title: Surgery for Locally Unresectable Pancreatic Cancer
Acronym: ROBIN
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Chief of General Surgery 2 Department - HBP and liver transplantion unit, Azienda Ospedaliera di Padova
Other Study IDs: AOP3371; 6096/AO/24 (Other: CET area centro-est Veneto)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
Keywords: Pancreatic cancer; Coversion Surgery Pancreatic Cancer; Quality of Life; Locally advanced PDAC; Unresectable Pancreatic Cancer; Neoadjuvant therapy for pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Each enrolled patient will complete quality of life questionnaires, specifically the EORTC QLQ-C30, PAN26, and EQ-5D, at different time points: at enrollment and every 2-3 months after surgery, for up to 2 years.

SUMMARY:
Pancreatic cancer is a severe disease often diagnosed at an advanced stage, when surgery is not possible. New chemotherapy treatments can sometimes shrink the tumor and make surgery an option. This study aims to understand if surgery after such treatments can improve survival and quality of life in selected patients treated at expert centers.

DETAILED DESCRIPTION:
Pancreatic cancer (PC) has a rising incidence and remains associated with one of the mostchallenging prognosis in oncology, with a 5-years survival around 11% and merely 4% of patients alive at 10 years. About one third of PC patients is diagnosed with locally advanced (LAPC) stage of disease, with a primary tumor that is considered unresectable (in the absence of metastatic disease) due to the local involvement of major vessels and is typically treated with palliative chemotherapy or best supportive care, with the aim to prolong survival while maintaining acceptable quality of life (QoL). However, the introduction of novel induction chemotherapy regimens has improved the clinical outcome of these patients in recent years. The preferred induction regimen for patients with favorable performance status (ECOG 0-1) has become modified 5-fluorouracil, leucovorin, irinotecan, and oxaliplatin [(m)FOLFIRINOX], with gemcitabine + nab-paclitaxel (GEMNabP) as a more tolerable alternative. In this scenario, the resection of apparently unresectable PC following induction chemotherapy, although somewhat controversial, has emerged as an important development for selected patients. In this regard, the National Comprehensive Cancer Network (NCCN) guidelines recommends 4 to 6 months of induction combination chemotherapy followed by conventional radiotherapy (CRT) or stereotactic body radiation therapy (SBRT) for selected patients without systemic metastases, followed by consideration for surgical resection if feasible, with adjuvant chemotherapy if clinically indicated. Surgical resection can be usually achieved in about 25% of LAPC patients after chemotherapy with modern regimens, and in the context of multidisciplinary management at high-volume centers with high expertise. Resection is associated with encouraging results in terms of median overall survival (OS), reaching 20 to 40 months, and with 5-years survival around 20%. To achieve surgical radicality, venous resection, arterial divestment or even arterial resection could be necessary. In recent multicentric series, patients receiving R0 portal vein (PV)/superior mesenteric vein (SMV) resection had a median OS of 24 months and a 20% 5-year OS 16, and patients requiring major arterial reconstruction and/or periarterial divestment had in-hospital mortality rates of 4-5%, median OS of 13.7-20.1 months, and 5-year OS of 12.5-13.7%. Despite the encouraging survival outcomes, based on both remarkable advances in surgical technique at high-volume centers and the use of modern combination chemotherapy regimens and chemo-radiation, aggressive surgery for LAPC after induction chemotherapy remains a controversial topic for several aspects:

* Most of the available literature consists of retrospective studies, without intention-to-treat design and with clear selection bias for best responders after induction therapy, who are selected for surgery. Other studies reported similar survival outcomes in non-resected LAPC patients who had a good radiographic and serologic response after first line chemotherapy. While standard dose RT appeared ineffective in patients who have not undergone resection, RT with dose intensification and ablative intent might enable improvements in local control in LAPC patients, and SBRT seems to successfully achieve local control while also improving QoL.
* Most series considered locally advanced and borderline resectable PC as a single entity or did not distinguish between arterial resection of common hepatic artery (CHA)/celiac trunk (CA) or superior mesenteric artery (SMA), despite clear differences in terms of prognosis and perioperative complexity. Surgery for LAPC is feasible and safe only at high-volume centers with dedicated programs, and arterial resections are technically demanding procedures with a long learning curve (esteemed around 15 procedures).
* Quality of life (QoL) and patient reported outcomes (PROMS) were seldom verified and put in the context of the relatively modest survival of resected LAPC patients. Despite improvements in recent years, arterial divestment or resections may not only increase significantly perioperative morbidity and mortality, but also imply life-long consequences such as diarrhea, due to nerve plexus dissection, and diabetes, as total pancreatectomy is often required. Despite its technical complexity, there is no high-level evidence supporting the benefit of aggressive surgery for LAPC after induction chemotherapy.

The aim of the present study is to evaluate survival and QoL outcomes in a cohort of patients affected by LAPC and selected for surgical exploration and radical resection after disease non progression during induction chemotherapy at leading expert centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients able to give informed consent
* Histologically confirmed pancreatic adenocarcinoma
* LAPC stage according to NCCN10 at diagnosis (Figure 1)
* Received at least 4 months of induction chemotherapy
* RECIST 1.1 stable disease (SD) or partial response (PR) after induction therapy
* Patient considered eligible for radical resection by local MDT

Exclusion Criteria:

* Informed consent withdrawal
* Presence of tumor characteristics precluding surgery
* Presence of patient significant comorbidities precluding surgery
* Unavailable pre-induction therapy abdominal imaging
* Pathological confirmation of any tumor different from PDAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with hystologically proved locally advanced pancreatic adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
HRQoL deterioration-free survival | From enrollment to the end of study period, set at 2 years
  The primary outcome is HRQoL deterioration-free survival, defined as the time from surgery until definite HRQoL score deterioration and including death from any cause as an event.

SECONDARY OUTCOMES:
Disease-specific survival (DSS) | 2 year from enrollment
Recurrence-free survival (RFS) | 2 year from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Chirurgia Generale 2, Azienda Ospedale di Padova, Padova, Italy 35128, Padua, Italy

IPD SHARING:
Plan to Share IPD: No